CLINICAL TRIAL: NCT03587779
Title: Comparison of the Effect of Sevoflurane and Desflurane on Patient State Index: A Randomized Controlled Trial
Brief Title: Comparison of Effect of Equi-MAC Anesthetics on PSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoung-Ho Ryu, MD, Assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-05-045
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia
Keywords: patient state index; sevoflurane; desflurane; minimum alveolar concentration
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia is maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia is maintained with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Throughout the study period, anesthesia is maintained with sevoflurane of age-corrected equivalent minimum alveolar concentration.
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Desflurane — Throughout the study period, anesthesia is maintained with desflurane of age-corrected equivalent minimum alveolar concentration.
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
The aim of this study is to compare the patient state index values produced by equi-MAC of sevoflurane and desflurane in patients undergoing single-agent volatile anesthesia.

DETAILED DESCRIPTION:
There have been several studies comparing electroencephalogram-derived indices produced by sevoflurane and desflurane. However, to the best of our knowledge, there has been no study which compared the two inhaled anesthetics using patient state index. Therefore, the aim of this study is to compare the patient state index values produced by sevoflurane and desflurane at equi-MAC in patients undergoing single-agent inhalation anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 19 and 65 yr
* patients with American Society of Anesthesiologists physical status classification I or II
* patients scheduled for elective surgery under volatile anesthesia
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any psychiatric or neurological disease
* patients receiving any medication affecting the autonomic or central nervous system
* patients with a history of alcohol or drug abuse
* pregnant or lactating women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
patient state index | After a 30-min waiting period from the induction of anesthesia
  patient state index value at a steady-state anesthesia of equi-MAC

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung-Ho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No